CLINICAL TRIAL: NCT05954611
Title: A Phase I, Randomized, Blinding, Single-dose, Placebo Control Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics Effect of GR2002 in Chinese Health Volunteers
Brief Title: The Study of Single Dose Administration of GR2002 Injection in Chinese Health Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genrix (Shanghai) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GR2002-001
Record Dates: First submitted 2023-05-26; First posted 2023-07-20 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GR2002 injection (Experimental): GR2002 subcutaneous injection
  Interventions: Biological: GR2002 injection
- placebo (Placebo Comparator): placebo subcutaneous injection
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: GR2002 injection — one single dose of GR2002 injection
  Arms: GR2002 injection
Biological: Placebo — one single dose of placebo
  Arms: placebo

SUMMARY:
To evaluate the pharmacokinetic (PK) characteristics and pharmacological effect of GR2002 injection in Chinese healthy volunteers

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled phase I clinical trial to evaluate the safety, tolerability, pharmacokinetics, preliminary pharmacodynamics, and immunogenicity characteristics of single subcutaneous administration of GR2002 injection in healthy adult Chinese subjects.

The initial dose group is 35mg, and the subsequent doses will gradually increase. Only after all subjects in the current dose group have completed at least 2 weeks of safety and tolerance observation and confirmed safe tolerance, can they enter the next dose group for medication observation until the "dose increase termination standard" is reached.

Follow up will be conducted for at least 12 weeks ± 3 days after completion of medication administration.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age of 18 to 55 years, inclusive, male or female 2. BMI between 19 kg/m2 and 26 kg/m2 (inclusive) 3. Healthy volunteers

Exclusion Criteria:

* 1. History of chronic disease or serious disease 2. Subject with severe psychological or mental illness 3. Not enough washing-out period for previous therapy 4. Other.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AE) | 85 days
  Incidence of AEs, including any abnormal physical examinations, abnormal vital signs, abnormal ECG, and abnormal lab testing

SECONDARY OUTCOMES:
Pharmacokinetics (PK) parameter: Time to reach peak concentration (Tmax) | 85 days
  Time to reach peak concentration (Tmax)
Pharmacokinetics (PK) parameter : Peak Plasma concentration (Cmax) | 85 days
  Peak Plasma concentration (Cmax)
Pharmacodynamics (PD): Changes from baseline in serum thymus activation regulation chemokine (TARC) concentration after GR2002 administration | 85 days
  Changes from baseline in serum thymus activation regulation chemokine (TARC) concentration after GR2002 administration
Immunogenicity: anti-drug antibody (ADA) and neutralizing antibody (Nab) | 85 days
  Detection of anti-drug antibody (ADA) and neutralizing antibody (Nab)

CONTACTS AND LOCATIONS:
Overall Officials: Yi Fang, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No